CLINICAL TRIAL: NCT00013091
Title: Treatment of Depression in Patients With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Masking: Single | Purpose: Treatment
Other Study IDs: IIR 95-074
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2009-05

CONDITIONS: PTSD; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Self-management therapy; Psychoeducational group therapy

INTERVENTIONS:
Behavioral: Self-management therapy; Psychoeducational group therapy

SUMMARY:
Post-traumatic stress disorder is a mental health problem of enormous proportion within the VA system for both male and female veterans. The 40 percent of veterans with PTSD and concurrent clinically significant depression are particularly difficult to treat. Effective and efficient treatment of veterans with this combination of disorders would be of benefit to a significant number of veterans.

DETAILED DESCRIPTION:
Background:

Post-traumatic stress disorder is a mental health problem of enormous proportion within the VA system for both male and female veterans. The 40 percent of veterans with PTSD and concurrent clinically significant depression are particularly difficult to treat. Effective and efficient treatment of veterans with this combination of disorders would be of benefit to a significant number of veterans.

Objectives:

Well-validated treatments of PTSD and its complications are rare. There are no studies of treatment addressing the sequelae of chronic PTSD, including depressive symptomatology. Our study is the first randomized, controlled study of group psychosocial interventions for the combination of PTSD and depression in male and female veterans. The purpose of the study is to evaluate the impact of two psychosocial interventions on clinical outcomes and on the use of hospital resources by veterans with these co-existing disorders.

Methods:

Male and female veterans with both PTSD and depressive diagnoses will be recruited for the study. Male veterans must have combat-related PTSD, and female veterans will have trauma related to sexual assault. Veterans will be randomly assigned to either Self-Management Therapy (Rehm, 1984), a cognitive-behavioral treatment program for depression, or to a Psychoeducational Group Therapy (Dunn, et al., 1998). Both programs involve short-term group therapies that teach veterans about their disorders, and provide them with new strategies and skills for overcoming them. These therapy groups will be in addition to other standard care that veterans receive within the Trauma Recovery Program at the Houston VA Medical Center. Approximately 120 male veterans and 60 female veterans will be enrolled in the program. Participants will be assessed at pretest, posttest, and at 3-, 6-, and 12-month follow-up periods, utilizing various clinician-administered and self-report instruments of psychiatric symptomatology, psychosocial functioning, constructs targeted by the therapy groups, treatment compliances, and satisfaction.

Status:

Final report preparation.

ELIGIBILITY:
Inclusion Criteria:

To be accepted in the study, patients must (a) meet criteria for combat-related (men's cohort) PTSD and either major depressive disorder of dysthymic disorder, (b) not meet criteria for current or past psychosis, score 24 or greater on a Mini-Mental State Examination cognitive screen, (d) not exhibit active suicidality or severity that would preclude participation in the groups, and (e) agree to random assignment and sign informed consent forms. For the women's groups, patients have PTSD related to sexual trauma.

Exclusion Criteria:

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 1997-10; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Jo Dunn, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

REFERENCES:
- [Result] Dunn NJ, Yanasak E, Schillaci J, Simotas S, Rehm LP, Souchek J, Menke T, Ashton C, Hamilton JD. Personality disorders in veterans with posttraumatic stress disorder and depression. J Trauma Stress. 2004 Feb;17(1):75-82. doi: 10.1023/B:JOTS.0000014680.54051.50. PMID 15027797